CLINICAL TRIAL: NCT03888703
Title: Early Intervention of Fractional Ablative CO2 Laser With or Without 830 nm LED Phototherapy for Acute Burn Injuries
Brief Title: The Use of Fractional Ablative CO2 Laser vs Control on Acute Traumatic Injuries to Prevent Scar Formation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Miami Dermatology and Laser Institute (Other)
Collaborators: CynosureLutronic (Industry)
Responsible Party: Principal Investigator, Jill Waibel, Owner of Miami Dermatology and Laser Institute, Board Certified Dermatologist, Director of Clinical Operations, Miami Dermatology and Laser Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SAIRB-13-0045
Record Dates: First submitted 2019-03-06; First posted 2019-03-25 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Scar; Trauma Injury; Burns; Wound Heal; Early Medical Intervention; Laser Therapy
Keywords: early laser intervention; scar prevention; laser resurfacing; wound healing
MeSH Terms: conditions — Cicatrix; Accidental Injuries; Burns

STUDY DESIGN:
Intervention Model Description: Each subject possessed extensive burn wounds. Wounds on each subject were divided into treatment arms of intervention with fractional ablative CO2 laser and control.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The treatment and control areas were randomized in advanced such that the investigator did not choose which sections to treat. Control areas were covered during the treatment so the investigator/provider could only see areas to be treated. Outcomes assessors evaluated photographs without knowledge of the identity of each area. The participant could not be masked due the experience of receiving treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Treatment (Experimental)
  Interventions: Device: Fractional ablative CO2 laser
- Control (No Intervention)

INTERVENTIONS:
Device: Fractional ablative CO2 laser — Three treatments with a fractional ablative CO2 laser 8 weeks apart
  Arms: Treatment

SUMMARY:
Surgical standard for treating traumatic burn injury scarring is to wait one year following the initial assault prior to beginning treatment. This study investigates the use of fractional ablative CO2 laser when begun within 3 months of a traumatic burn injury and it's impact on scar formation compared to the control. We hypothesized that early intervention would substantially mitigate the formation of scar tissue and help restore more normal appearing skin.

ELIGIBILITY:
Inclusion Criteria:

* Subject is between 18 and 80 years of age with burn injuries suffered within the prior 3 months
* Subject is a healthy Male or Female
* Fitzpatrick Skin Type I - IV
* Subject must have moderate - severe burn damage of sufficient bilateral area involving either the face, trunk, arms or legs
* Subject must be able to read, understand and sign the Informed Consent Form
* Subject must be willing and able to adhere to the treatment and follow-up schedule and post-treatment care instructions
* Subject must be willing to have limited sun exposure for the duration of the study, including the follow-up period
* Subject is willing to have photographs taken of the treated area which will be used de-identified in evaluations and may be used de-identified in presentations and/or publications
* For female candidates - they may be post-menopausal, surgically sterilized, or using a medically acceptable form of birth control during the entire course of the study.
* Female candidates with child bearing potential - willing to take pregnancy test and result must be negative.

Exclusion Criteria:

* Subject is less than 18 or greater than 80 years of age.
* Subject has Fitzpatrick Skin Type V - VI
* Subject is Pregnant or planning to become pregnant during the study duration
* Subject is breast feeding during the study duration
* Subject has an active skin infection, dermatitis or a rash in the treatment area
* Subject has a history of immunosuppression/immune deficiency disorders or currently using immunosuppressive medications
* Subject has a known bleeding disorder
* Subject has a known photosensitivity to the study laser wavelength, history of ingesting medications known to induce photosensitivity, or history of seizure disorders due to light.
* Subject has a known collagen, vascular disease or scleroderma
* Subject has undergone any surgery or other procedures in the treatment area within 6 months of treatment which are still healing.
* Subject is suffering from significant concurrent illness, such as insulin-dependent diabetes, peripheral vascular disease or peripheral neuropathy
* Subject is undergoing systemic chemotherapy for the treatment of cancer
* Subject has lesions suspicious for malignancy
* The systemic use of isotretinoin (Accutane®) or other retinoid derivatives within 6 months of study participation
* Any use of gold therapy for disorders such as rheumatologic disease or lupus
* The subject is excessively tanned in areas to be treated or unable/unlikely to refrain from tanning during the study
* The subject has participated in a study of another device or drug within three months prior to enrollment or during the study.
* As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-05-04 (Actual); Primary Completion 2017-05-05 (Actual); Study Completion 2017-05-05 (Actual)

PRIMARY OUTCOMES:
Manchester Scar Scale | From the day of the first treatment prior to intervention and at 6 months following the final treatment
  The sum total of the Manchester Scar Scale to assess the change in scar characteristics. The scale includes the following categories: Color, matte vs shiny, contour, distortion, and texture. Scales for color, contour, distortion, and texture are rated on a 1-4 scale with 1 being most normal and 4 being most abnormal. Matte vs shiny is rated on a 1 to 2 scale with 1 being matte and 2 being shiny. Assessments completed by blinded evaluators. A decrease in score indicates improvement in scar characteristics.
Digital photography | From the day of the first treatment prior to intervention and at 6 months following the final treatment
  Visual improvement as demonstrated in digital photography. Before and after photos identified by blinded evaluators
Changes in scar characteristics such as dermal and epidermal character as well as vascular structure and organization assessed through histology. | From the day of the first treatment prior to intervention and at 6 months following the final treatment
  Some patients elected to do optional biopsies for deeper evaluation of changes in skin structure. Biopsies were taken prior to treatment and 6 months following treatment to assess dermal and epidermal character as well as the size and organization of vasculature. Evaluation was done qualitatively.

SECONDARY OUTCOMES:
Optical Coherence Tomography | From the day of the first treatment prior to intervention and at 6 months following the final treatment
  Patients were scanned using OCT for noninvasive skin imaging of both control and treatment areas
Treatment Time | Treatment time was measured at each of the three treatments conducted on day 0, day 60, and day 120
  The total duration of each treatment was measured in minutes to assess treatment characteristics for large surface areas
Severity of post treatment cutaneous responses as evaluated by the investigator | Post treatment response was assessed immediately post treatment at each of the three treatments conducted on day 0, day 60, and day 120
  Cutaneous responses including purpura, edema, erythema, hyperpigmentation, hypopigmentation, blistering and scarring were assessed following each treatment. Areas were rated on a 1-4 scale where 1 = none, 2 = mild, 3 = moderate, and 4 = severe.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Waibel JS, Gianatasio C, Rudnick A. Randomized, Controlled Early Intervention of Dynamic Mode Fractional Ablative CO2 Laser on Acute Burn Injuries for Prevention of Pathological Scarring. Lasers Surg Med. 2020 Feb;52(2):117-124. doi: 10.1002/lsm.23170. Epub 2019 Oct 20. PMID 31631361